CLINICAL TRIAL: NCT06109701
Title: Efficacy of Air-polishing on Pain Perception and Compliance Rate to Periodontal/Peri-implant Maintenance Therapy: a 2-year Follow-up Randomized Controlled Clinical Trial
Brief Title: Efficacy of Air-polishing on Pain Perception and Compliance Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Tiago Ribeiro Amaral, PhD candidate, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PER-ECL-2021-08
Record Dates: First submitted 2023-09-06; First posted 2023-10-31 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis
Keywords: Peri-implantitis; prevention; peri-implant mucositis; pain perception
MeSH Terms: conditions — Peri-Implantitis | interventions — Debridement; Tooth Exfoliation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group - Ultrassonic Devices (Active Comparator): Supra and sub-gingival debridement with an ultrasonic device (DTE-D5, Woodpecker®, Guilin, China) with a plastic tip (Hu-Friedy®, Rockwell St, Chicago, IL, USA) and scaling with plastic curettes (Hu-Friedy®, Rockwell St, Chicago, IL, USA) around dental implants and a conventional metal tip for teeth will be used.
  Interventions: Procedure: Debridement with ultrasonic device and scaling with plastic curettes
- Test Group - Erythritol based air-polishing powder (Experimental): Supra and sub-gingival debridement with an erythritol based air-polishing powder (Air-Flow, EMS, Nyon, CH) will be used during 5 seconds on each site (Schwarz et al., 2015).
  Interventions: Procedure: Debridement with erythritol based air-polishing powde

INTERVENTIONS:
Procedure: Debridement with ultrasonic device and scaling with plastic curettes — Supragingival and subgingival debridement
  Other Names: Supportive periodontal / peri-implant treatment
  Arms: Control Group - Ultrassonic Devices
Procedure: Debridement with erythritol based air-polishing powde — Supragingival and subgingival debridement
  Other Names: Supportive periodontal / peri-implant treatment
  Arms: Test Group - Erythritol based air-polishing powder

SUMMARY:
Implants have become a popular and widely used treatment option for treating partial and total edentulism. As the number of implants placed increases, so does the incidence of peri-implant mucositis and peri-implantitis. Placing patients under SPT/maintenance care has been shown to prevent and treat such conditions. Despite SPT's importance in prevention and infection control, adherence to scheduled SPT visits have been unsatisfactory. Understanding the reasons for non-compliance can help both the clinician and research community to address them by improving patients experience to those visits thereby increasing compliance.

DETAILED DESCRIPTION:
Objectives:

1. General objective Evaluate the patient reported outcomes to a different implant instrumentation method during SPT visits, as well as its effect in compliance rates and clinical outcomes.
2. Specific objective

   1. To evaluate pain/discomfort during SPT around dental implants and teeth.
   2. To evaluate pain/discomfort during SPT around healthy and diseased dental implants.
   3. To evaluate patient reported outcomes and clinical variables by decontamination during SPT with erythritol based air polishing powder (Air Flow Master, Air-Flow Plus, EMS, Nyon, Switzerland), at the first SPT, at 1 and 2 years.
   4. To evaluate the effect of erythritol based air polishing powder (Air Flow Master, Air-Flow Plus, EMS, Nyon, Switzerland) during SPT on the compliance rates after 1 and 2 years of follow-up.
   5. Hypothesis:

a) General Hypothesis The proposed protocols, focused on the prevention of peri-implantitis, will result in an increase adherence to SPT by better understanding the specific factors related to non-compliance, specifically by improving the experience of patients to SPT visits.

b) Specific Hypothesis

1. SPT with conventional ultrasonic device will result in more pain/discomfort around dental implants than in teeth.
2. SPT by means of an erythritol based air-polishing powder (Air Flow Master, Air-Flow Plus, EMS, Nyon, Switzerland) will result in better patient reported outcomes and same clinical outcomes, at the first SPT and after 2 years.
3. SPT by means of an erythritol based air-polishing powder (Air Flow Master, Air-Flow Plus, EMS, Nyon, Switzerland) will result in the increase of the compliance rates after 2 year of follow-up.

6. Material y Methods: Study Design The present research project is designed as a randomized controlled clinical trial with a 2-year follow-up. The reporting of this clinical trial will follow the Consolidated Standards of Reporting (CONSORT) guidelines.

Subject Selection The study will be performed after the approval of the Ethics Committee of the Universitat Internacional de Catalunya (UIC) and will be conducted according to the principles outlined in the Declaration of Helsinki and Ethical Conduct for Research with Human Beings.

A list of patients who have been enrolled in SPT at the Department of Periodontology of UIC and met the inclusion criteria will be used - patients will be called once every 2 days (with a maximum of 3 attempts) for a SPT visit by the same investigator (E.R).

- SPT visit One calibrated investigator will consecutively call patients for SPT visits and will be responsible of enrolling the patients (E.R).

The study variables will be recorded in a case report form (CRF) specially designed for the study. Each study patient will be assigned a numerical code comprising a 3-digit patient code (assigned correlatively as they are included in the study). Only the study investigator will be able to identify the patient by their code.

Screening examination The clinician will review with the patient the Information and Medication History Forms and record the anthropometric, socio-demographic and clinical information. Candidates will undergo an oral pathology examination and a full-mouth manual probing using a periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) to determine their periodontal and peri-implant status. Presence or absence of plaque will be recorded after staining with an erythrosine disclosing dye (Plac-Control®, Dentaid SL, Cerdanyola, Spain). Finally, periapical radiographs (Dürr Dental AG, Bietigheim-Bissingen, Germany) of all implants will be taken using a paralleling cone technique and a film-holder (7mA- 60kV/20ms).

The same calibrated examiner (E.R) will record clinical variables of mPI, BOP, PPD, MR and clinical attachment level (CAL).

Randomization and study groups Once oral hygiene instructions were provided, patients will be randomly assigned to the Test or Control groups. Allocation of patients will be decided following randomization tables with permuted blocks of four while the information will be concealed by using opaque envelopes, which will be labelled with the patient study number and only be revealed after oral hygiene instructions are provided.

Questionnaires A blinded calibrated examiner (C.V) will give each patient the following questionnaires.

Pain Perception Pain experienced during the SPT visit will be recorded using the Visual Analog Scale (VAS). A horizontal 10 cm VAS (graded from zero, representing no pain, to 10, representing the worst pain possible) will be used by the patients immediately after finishing the supragingival debridement around teeth, and then, after performing supragingival debridement around the dental implants.

Modified Dental Anxiety Scale (MDAS) Another questionnaire (MDAS) will be used to measure patient anxiety towards SPT visit in both groups. The MDAS consists of five questions answered with a 5-category Likert scale, ranging from 'not anxious' to 'extremely anxious'. The original MDAS questionnaire does not cover anxiety toward SPT visits. Therefore, a question enquiring about patients' feelings toward SPT visit will be added. Patients will complete the modified MDAS once, after finishing the SPT visit.

- Follow-up SPT visits Patients enrolled in the study will be called for SPT every 4 months (to standardize every patient during the time of the study) and supragingival debridement will be performed accordingly to their group (control or test). All clinical and microbiological variables will be re-examined by the same blinded examiner (E.R) after the first SPT visit (4 months), at 1 year and 2 years of follow-up. Additionally, a periapical radiograph of all implants involved in the study will be taken at 1 year and 2 years of follow-up. Individual compliance will be registered as well in the CRF.

Patients will be further motivated with respect to oral hygiene habits during the entire period of the study.

Clinical examination A guidebook will be prepared to standardize procedures throughout the protocol, step by step, for all questionnaires and evidence collection. The data will be transferred to a computerized database.

The study variables will be recorded in a case report form (CRF) specially designed for the study. Each study patient will be assigned a numerical code comprising a 3-digit patient code (assigned correlatively as they are included in the study). Only the study investigator will be able to identify the patient by their code.

Determination of recurrent sites and re-treatment needs Sites will be determined as re-treatment needs if they show PD ≥ 4 mm and CAL ≥ 4 mm in more than 2 non-adjacent teeth, together with the presence ≥10% of BOP and/or SU (around teeth) and if they show PD ≥ 6mm, together with BOP and/or SU, and bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant (around dental implants), during SPT appointment. Individuals will be treated with non-surgical or surgical procedures, where necessary, by postgraduate students of the Periodontology Department at the CUO (UIC).

Intra-examiner reproducibility Reproducibility of clinical examinations will be conducted by the examiner (E.R), evaluating the Implant PPD and mBI in 5 patients, not involved in the study, on two separate occasions, 1 week apart. The intra-class correlation coefficient and the kappa index will be calculated. Calibration will be accepted when measurements at baseline and at one-week evaluation will be within a difference of 0.5 mm >90% of the time.

Withdrawal of consent The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation. Such withdrawal will be documented in the medical record file. Losses to follow-up are taken into account in the sample size calculations (12%).

Statistical analysis Descriptive analysis Descriptive statistical methods (percentage and numbers on total) will be used to analyze the evaluated parameter Inferential analysis Data will be calculated at patient level and implant/tooth level. VAS score will be considered as the main outcome (quantitative).

If the distribution is normal, the following tests will be used:

* Binary categorical variables: T-Student / Fisher's exact test;
* Categorical variables with > 2 categories: ANOVA;
* Quantitative variables: Simple linear regression / Pearson correlation coefficient.

If it doesn't follow normality:

* Binary categorical variables: U of Mann-Whitney;
* Categorical variables> 2 categories: H of Kruskal-Wallis;

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients, rehabilitated with at least one dental implant in the maxilla or mandible with at least 3 years of function;
* No implant mobility;
* Treated periodontal disease;
* Non-smoker or light smoking status in smokers (<10 cigarettes/day).

Exclusion Criteria:

* Patients with diagnosed fibromyalgia disorder or who are taking drugs that might influence the perception of pain (i.e., opioids, gabapentin) will be excluded from the study (Alcalde et al. 2017).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Pain/Discomfort (VAS) reported after decontamination during SPT. | immediately after the procedure
  0 = no pain and 10 = extreme, unbearable pain

SECONDARY OUTCOMES:
Compliance to Supportive Periodontal Treatment (SPT) reported after decontamination during SPT. | 24 months
  Regular Complier = 3- to 6-month recall interval (≥2 SPT/year) Erratic Complier = 7- to 12-month recall interval (<2 SPT/year) Non-Complier = no recall interval program (no SPT/year)
Changes in Full mouth plaque index (FMPI) | 24 months
  Full mouth plaque index (FMPI) will be assessed dichotomously at four sites per tooth (mesial, buccal, distal and lingual). Presence or absence will be recorded after staining with an erythrosine disclosing dye (Plac-Control®, Dentaid SL, Cerdanyola, Spain). Presence of plaque will be scored if an area of clearly stained material is present along the gingival margin and if this material can be removed with the side of the probe. The percentage of surfaces with plaque out of the total number of examined tooth surfaces will be calculated
Changes in Full mouth plaque index (FMBI) | 24 months
  Full mouth bleeding index (FMBI) will be assessed dichotomously as presence or absence of bleeding after 30 seconds of gently probing. The proportion of bleeding surfaces out of the total number of examined surfaces will be calculated (Ainamo and Bay, 1975).
Changes in Periodontal probing depth (PPD) | 24 months
  Full mouth PPD measured at six aspects around tooth.
Changes in gingival recession (GR) | 24 months
  Gingival Recession (GR) will be recorded at six aspects per implant: mesial buccal, buccal, disto-buccal, mesio-lingual, lingual and disto-lingual.
Changes in modified Plaque Index (mPI) | 24 months
  mPI will be measured at six aspects around implants: Score 0 - no detection of plaque. Score 1 - plaque only recognized by running a probe across the smooth marginal surface of the implant.
  Score 2 - plaque can be seen by the naked eye. Score 3 - abundance of soft matter.
Changes in modified Bleeding Index (mBI) | 24 months
  mBI will be assessed 30 seconds after 0.15 N force probing. Score 0 - no bleeding. Score 1 - isolated bleeding spots visible. Score 2 - blood forms a confluent red line on margin. Score 3 - heavy or profuse bleeding. This variable will be dichotomized in presence/absence of bleeding and will serve as the main variable.
Changes in suppuration on probing (SOP) | 24 months
  SOP evaluated after assessing dichotomously the presence of suppuration within 30 seconds after gentle probing.
Changes in Implants probing depth (implant PPD) | 24 months
  Implant PPD, measured from the mucosal margin to the bottom of the probable pocket, determined at six aspects per implant: mesial-buccal, buccal, disto-buccal, mesial-lingual, lingual and disto-lingual with a resin splint.
Changes in Mucosal Recession (MR) around dental implants | 24 months
  MR at dental implants will be recorded at six aspects per implant: mesial-buccal, buccal, disto-buccal, mesial-lingual, lingual and disto-lingual.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina V Vallès, Dentist, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Clínica Universitaria de Odontologia, Sant Cugat del Vallès, Barcelona, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06109701/Prot_SAP_000.pdf